CLINICAL TRIAL: NCT06924255
Title: An 8-week Open-label, Multicenter Randomized Study of Accelerated and Slower Switching to Xanomeline/Trospium Following Atypical Antipsychotic Treatment to Assess the Safety, Tolerability, and Efficacy in Participants With DSM-5 Schizophrenia
Brief Title: An 8-week Open-label Study of an Accelerated and Slower Switching to Xanomeline/Trospium Following Atypical Antipsychotic Treatment in Participants With Schizophrenia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Collaborative Neuroscience Research, LLC (Network)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0079
Record Dates: First submitted 2025-03-31; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia Disorders
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- accelerated transition (Other): accelerated transition arm will reduce the atypical AP treatment at a rate of 50% of the initial treatment over a 2-week period,
  Interventions: Drug: Xanomeline and Trospium Chloride
- slower transition (Other): slower transition arm will reduce the atypical AP treatment at a rate of 25% of the initial treatment over a 4-week period
  Interventions: Drug: Xanomeline and Trospium Chloride

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride — accelerated titration of Xanomeline and Trospium Chloride
Drug: Xanomeline and Trospium Chloride — slow titration of Xanomeline and Trospium Chloride

SUMMARY:
The study design is a de-escalation of current atypical AP treatment to X/T at a maintenance dose of X/T established either at 100 mg xanomeline/20 mg trospium chloride BID (total daily dose 200 mg xanomeline/40 mg trospium chloride) or 125 mg xanomeline/30 mg trospium chloride BID (total daily dose 250 mg xanomeline/60 mg trospium chloride) based on participants' clinical response and/or tolerability. While the package insert for X/T provides guidance for clinicians on dosing, this study is designed to assess how transitioning will occur in the "real world" situation.

DETAILED DESCRIPTION:
This will be a 2-arm, multicenter, randomized, 8-week, open-label study to evaluate the safety and tolerability, as well as the efficacy, of transition in adult participants with schizophrenia in an outpatient setting from oral atypical AP treatment to X/T.

The study design is a de-escalation of current oral atypical AP therapy to a X/T via accelerated or slower transition from current treatment.

The study will consist of a Screening Phase of up to 14 days, a Pre-switch Baseline Visit, an 8 week open-label Treatment Phase, and a safety Follow-up/End of Study (EOS) Visit at 7+2 days following the last dose of X/T for participants who complete the Treatment Phase and those who prematurely discontinue from the study. Participants who prematurely discontinue from the study due to AEs or lack of efficacy will be encouraged to continue with study procedures even though they are no longer receiving study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged 18 to 65 years, inclusive, at Screening.
2. Participant is capable of providing informed consent.

   1. A signed informed consent form (ICF) must be provided before any study assessments are performed.
   2. Participant must be fluent in English (oral and written) as the language of the ICF to consent. No translations will be permitted.
3. Participant has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (American Psychiatric Association 2013) criteria and confirmed by MINI for Schizophrenia and Psychotic Disorder Studies version 7.0.2.
4. Participant has not required psychiatric hospitalization, acute crisis intervention, or other increase in level of care due to symptom exacerbation within 12 weeks of Screening and is psychiatrically stable in the opinion of the Investigator.
5. PANSS Total Score of ≤80 at Screening and Baseline Visits.

   a. Score of ≤4 for the following core Positive Subscale items on PANSS: i. Item 2 (P2): Conceptual disorganization ii. Item 7 (P7): Hostility
6. CGI-S score of ≤4 at Screening and Baseline Visits.
7. Participant must be judged by the Investigator to be an appropriate candidate for transitioning from current oral AP medication due to safety or tolerability concerns and/or insufficient efficacy.
8. Participant is taking an oral AP and the AP regimen has been stable for at least 6 weeks prior to Screening. Participants are permitted to remain on non-prohibited (see Section 5.2, Exclusion Criterion #14, and Section 7.8) psychotropic medications (that are not secondary AP treatments) other than the primary pre-switch AP that have been part of their ongoing treatment regimen.

   1. For at least 6 weeks prior to Screening, the participant must be taking a single oral atypical AP medication at a dose and frequency consistent with the drug label. Low dose quetiapine (e.g., taken for sleep) taken in the 6 week prior to Screening is not exclusionary but must be discontinued by the Baseline Visit.
   2. Participant must be currently treated with one of the following selected atypical oral AP at the same dosing regimen at package insert specified dose range for schizophrenia for ≥6 weeks:

      * Risperidone
      * Paliperidone
      * Aripiprazole
      * Ziprasidone
      * Quetiapine
      * Lurasidone
      * Lumateperone
      * Brexpiprazole
      * Olanzapine No participants taking first-generation (typical) AP are to be included in the study.
9. In the opinion of the Investigator, it is clinically appropriate for the participant to discontinue current AP therapy and initiate treatment with X/T.
10. Participant is willing and able, in the opinion of the Investigator, to discontinue all secondary AP medications prior to Baseline visit.
11. BMI must be ≥18 and ≤40 kg/m2.
12. Participant resides in a stable living situation and is anticipated to remain in a stable living situation for the duration of study enrollment, in the opinion of the investigator.
13. Individuals of childbearing potential (IOCBP) must be willing and able to adhere to the contraception guidelines as defined in Appendix 1.

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 6 months before Screening (confirmed using MINI version 7.0.2 at Screening). Exclusionary disorders include, but are not limited to, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder, and posttraumatic stress disorder. Symptoms of mild mood dysphoria or anxiety are allowed as long as these symptoms are not the primary focus of treatment.
2. Participant has a history of moderate to severe alcohol use disorder or a substance (other than nicotine or caffeine) use disorder within the past 6 months or a positive urine drug screen (UDS) for a substance other than cannabis at Screening or Baseline.

   1. Participants with mild substance use disorder within the 6 months before Screening must be discussed and agreed upon with the Principal Investigator (PI) before they can be allowed into the study.
   2. Participants with positive UDS for cannabis are permitted to enroll in the study provided that the participants' pattern of use is not indicative of a substance use disorder.
   3. Urine toxicology screen positive for phencyclidine, amphetamines, opiates, cocaine, or alcohol (clinically significant alcohol use in the opinion of the Investigator).
3. History or presence of clinically significant cardiovascular (e.g., untreated or unstable hypertension, clinically significant tachycardia), pulmonary, renal, hematologic, gastrointestinal (GI, e.g., obstructive disorders [including conditions that may decrease GI motility, such as ulcerative colitis, intestinal atony, and myasthenia gravis], endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the participant or the validity of the study results.
4. Participant with cirrhosis, biliary duct abnormalities, and/or hepatobiliary carcinoma based on either medical history or liver function test results.
5. All grades of hepatic impairment (mild [Child-Pugh Class A], moderate [Child-Pugh Class B], and severe [Child-Pugh Class C]).
6. History or high risk of urinary retention or gastric retention.
7. History of narrow-angle glaucoma.
8. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months.
9. Risk for suicidal behavior during the study as determined by the Investigator's clinical assessment. Non-suicidal self-injurious behavior is not exclusionary.
10. Clinically significant abnormal finding on the physical examination, medical history, or clinical laboratory results at Screening.
11. An eGFR of < 60 mL/min
12. Elevations in hepatic transaminases at screening ≥3× ULN for ALT and AST and/or bilirubin > 2× ULN, unless in the context of Gilbert's syndrome
13. History of unstable hypertension or tachycardia as evidenced by:

    1. Blood pressure of ≥160/100 mmHg (single seated measure) at screening
    2. Heart rate of ≥110 bpm (single seated measure) at Screening
14. Participant is receiving other psychotropic medications for psychiatric and neurological conditions with Anticholinergic Risk Scale (ARS) scores >1 (tricyclic antidepressants, paroxetine, antispasmodics, antihistamines with anticholinergic properties).
15. History of treatment resistance to schizophrenia medications defined as:

    1. Failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) within the past 12 months OR
    2. Has a history of having received clozapine
16. Participant is receiving a long-acting injectable AP.
17. Developmental disorder, intellectual disability, or autism spectrum disorder (by history), with the exception of participants diagnosed with autism at age <18 due to historic diagnostic criteria precluding schizophrenia diagnoses of minors (at discretion of Investigator).
18. Lifetime history of clinically significant head trauma.
19. Pregnant, breastfeeding, or less than 3 months postpartum.
20. Active biliary disease (e.g., symptomatic gallstones). Participants with other biliary histories are eligible and should be discussed with the Medical Monitor.
21. Participants with any of the following:

    1. History of bladder stones
    2. History of recurrent urinary tract infections
    3. For male participants, serum prostate-specific antigen >10 ng/mL at Screening
    4. For male participants ≥45 years of age, International Prostate Symptom Score (IPSS) of 5 (i.e., "almost always") on items 1, 3, 5, or 6
    5. For male participants ≥45 years of age, an IPSS ≥9 for the sum of items 1, 3, 5, and 6
22. In the opinion of the Investigator (and/or Sponsor), participant is unsuitable for enrollment in the study, or participant has any finding that, in the opinion of the Investigator (and/or Sponsor), may compromise the safety of the participant or affect their ability to adhere to the protocol visit schedule or fulfill visit requirements.
23. Participant has had psychiatric hospitalization(s) for more than 30 days (cumulative) within the 12 months before Screening.
24. Participant with prior exposure to X/T or who has a history of prior X/T intolerability (allergy/hypersensitivity).
25. Risk of violent or destructive behavior in the opinion of the Investigator.
26. Current involuntary hospitalization or incarceration.
27. Participation in another clinical study in which the participant received an experimental or investigational drug agent within 3 months prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
discontinuation rate of accelerated and slower switching of atypical antipsychotic (AP) treatment to xanomeline and trospium chloride (X/T) | 8 weeks
  To evaluate all-cause X/T discontinuation rate of accelerated and slower switching of atypical antipsychotic (AP) treatment to xanomeline and trospium chloride (X/T) over a period of 8 weeks

SECONDARY OUTCOMES:
evaluate the effectiveness of switching outpatients from standard atypical AP treatment to X/T | 8 weeks
  To evaluate the effectiveness of switching outpatients from standard atypical AP treatment to X/T over a period of 8 weeks
evaluate the safety and tolerability of X/T following switch from atypical AP | 8 weeks
  To evaluate the safety and tolerability of X/T following switch from atypical AP

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - CenExel CIT LA, Bellflower, California
  - CenExel CNS - Garden Grove, Garden Grove, California
  - CenExel CIT IE, Riverside, California
  - CenExel CNS - Torrance, Torrance, California
  - CenExel RCA, Hollywood, Florida
  - CenExel CBH, Gaithersburg, Maryland
  - CenExel HRI Marlton, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided
Deciding on what journals to submit data